CLINICAL TRIAL: NCT04898127
Title: Antigen Rapid Test Screening to Prevent SARS-CoV-2 Transmission at Mass Gathering Events. A Randomised Trial.
Brief Title: Antigen Rapid Test Screening to Prevent SARS-CoV-2 Transmission (COVID-19) at Mass Gathering Events.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study needed approval from local authorities (City of Oslo and City of Bergen) to take place, which it did not get.
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CristinID2510078
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: COVID-19; Infection control; Rapid test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Individually randomised trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid test and concert (Experimental): Participants in this arm will be offered access to a concert, after a negative rapid test.
  Interventions: Diagnostic Test: SARS-CoV-2 antigen rapid test
- Control (No Intervention): Participants in this are will not be offered access to a concert during the study period.

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 antigen rapid test — Rapid test before access to mass gathering event (concert), provided the test result is negative.
  Arms: Rapid test and concert

SUMMARY:
To investigate the impact of rapid antigen testing for Severe Acute Respiratory Syndrome Corona Virus-2 (SARS-CoV-2), the investigators plan to conduct a large trial to assess the impact of using rapid tests to screen people before participating at a mass gathering event, i.e. a music concert. Among participants who wish to attend and fulfill the inclusion criteria, half will be offered access to rapid testing and concert (provided the test is negative), and the other half will not. Allocation will be by randomisation. A week after the concert both groups will be tested by means of a standard PCR-test.

DETAILED DESCRIPTION:
To investigate the impact of rapid SARS-CoV-2 antigen testing on the incidence of COVID-19, the investigators plan to conduct a large trial to assess the impact of using rapid tests to screen people before participating a mass gathering event, i.e. a music concert. The hypothesis is that screening by means of rapid testing eliminates any increase in risk of COVID-19 from attending a mass gathering event.

The investigators will recruit Individuals aged 18-45 years, who wish to attend a specific concert, have not received vaccination or had Covid-19 in the past six months, and are not in any risk group for severe disease. At recruitment, all participants (both concert and no-concert groups) will sign a consent form where they commit to using a contact tracing app, and to allowing the research group to use their data in the Norwegian Emergency Preparedness Register (BEREDT C19). They will also consent to having a COVID-19-test (PCR) conducted 6-8 days after the concert date.

After placing their payment, they will be randomised to be given access to a music concert (concert group), or not (no-concert group). Those who are randomised to the concert group will be tested for SARS-CoV-2 using a rapid antigen test, shortly before the concert. Those who test positive will be excluded from attending the concert and will immediately be offered a PCR-test.

All participants will be instructed to stay at home if they have symptoms of COVID-19 or are in quarantine. Participants who have symptoms or are quarantined at the time of the follow-up test will be offered a test through home visit by a mobile clinic.

Infection control measures will be applied to all concert participants in line with standards established by the sector, e.g. hand hygiene measures and a logistical system that seeks to minimise the risk of transmission during entry to the arena and exit after the concert

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years
* Willingness to be randomised and to have a PCR-test taken a week after mass gathering event (both intervention and control groups)

Exclusion Criteria:

* Vaccinated for COVID-19
* Having tested positive for SARS-CoV-2 the last 6 months
* Risk factors for severe COVID-19

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | 6-8 days after mass gathering event
  Positive PCR-test

SECONDARY OUTCOMES:
Clinical COVID-19 disease | 1 to 14 days after mass gathering event
  Registered diagnosis in administrative databases
Hospital admissions | 1 to 3 weeks after mass gathering event
  Registered in administrative database
False positive rapid test | Within 24 hours.
  Rapid tests that yield a positive result which is not confirmed by PCR test

CONTACTS AND LOCATIONS:
Overall Officials: Atle Fretheim, PhD, Principal Investigator — Norwegian Institute of Public Health

IPD SHARING:
Plan to Share IPD: Yes
We will collect very limited IPD: Beyond outcome measures, the IPD will be age, sex. These data can be shared, at the individual level.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Until 31. July 2026.